CLINICAL TRIAL: NCT00853229
Title: Pregabalin (Lyrica) for the Treatment of Vulvodynia: A Randomized, Double-blinded, Placebo-controlled Cross-over Study
Brief Title: Pregabalin for the Treatment of Vulvodynia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Not feasible due to low accrual
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: CCF 08-195
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Results first posted 2017-05-15 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Vulvodynia; Vulvar Vestibulitis
Keywords: vulvodynia; vulvar vestibulitis; chronic vulvar pain; generalized vulvodynia; localized vulvodynia
MeSH Terms: conditions — Vulvodynia; Vulvar Vestibulitis | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- pregabalin/placebo (Experimental): pregabalin and placebo given using a cross-over design
  Interventions: Drug: pregabalin
- placebo/pregabalin (Experimental): placebo and pregabalin given using a cross-over design
  Interventions: Drug: pregabalin

INTERVENTIONS:
Drug: pregabalin — pregabalin 150mg twice daily for 4 weeks
  Other Names: Lyrica

SUMMARY:
The purpose of this study is to determine whether pregabalin is effective in the treatment of vulvodynia.

DETAILED DESCRIPTION:
Vulvodynia is a condition exclusive to women and involves mostly burning, rawness, and itching of the external genitourinary tract that often results in painful intercourse. Vulvodynia rarely results in severe morbidity or mortality; rather it causes symptoms of the lower genital, urinary, and gastrointestinal tracts that can impact a woman's daily activities and negatively affect her quality of life.

Despite the fact that chronic vulvovaginal symptoms are one of the most common reasons for visits to a gynecology clinic, epidemiologic studies of the incidence and prevalence of these conditions are rare and available population-based studies are limited. Approximately 16% of women will experience chronic vulvar pain at some point in their lifetime; with 5% experiencing this condition before age 25.

Treatment approaches include behavioral changes, medical management, and surgery, specifically vulvar vestibulectomy. Prior to considering surgical intervention, all medical treatment options should be exhausted. Although vulvodynia is quite prevalent and can be a debilitating disease, there are few studies that critically evaluate the medical management of vulvodynia. Pregabalin is an anticonvulsant that has proven efficacy in the treatment of diabetic neuropathy, post-herpetic neuralgia, and fibromyalgia. Anecdotal data and one case report provide hope that this medication may also be effective in the treatment of vulvodynia.

ELIGIBILITY:
Inclusion Criteria:

* Adult women age 18 or greater
* Vulvodynia as defined as chronic vulvar discomfort or pain, characterized by burning, stinging, irritation or rawness of the female genitalia in cases in which there is no infection or skin disease of the vulva or vagina causing these symptoms. Pain may be constant or intermittent, localized or diffuse. Symptoms may be consistent with either Generalized Vulvodynia (diffuse or focal and constant or unremitting symptoms present in the labia majora, labia minora, and/or the vestibule that are not necessarily caused by touch or pressure to the vulva) or Vulvar Vestibulitis Syndrome (pain only in the vestibule and only during or after touch or pressure is applied).
* Pain ≥ 40 on 100mm VAS
* Practicing reliable form of birth control defined as sterilization, hormonal contraception, abstinence, IUD
* Must be able to attend follow up visits and are not likely to leave the area during the study period

Exclusion Criteria:

* Atrophic vaginitis, active bacterial vaginosis, yeast, and herpetic infections
* Current pregnancy diagnosed by positive serum or urine pregnancy test
* Current breastfeeding
* Seizure disorder or other chronic neurologic disease
* Diagnosis of chronic renal insufficiency defined as creatinine >1.4
* Unable to read and speak English
* Contraindication to pregabalin or history of prior use of pregablin
* Chronic narcotic or benzodiazepine use
* Chronic alcohol abuse
* Other chronic pain disorders, (ie. chronic pelvic pain, endometriosis, interstitial cystitis)
* Chronic neuropathic pain or anything affecting sensation (ie. MS, stroke)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-02; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beri M Ridgeway, MD, Principal Investigator — The Cleveland Clinic; Matthew D Barber, MD, MHS, Study Director — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Pregabalin First 4 Weeks: pregabalin and placebo given using a cross-over design
  pregabalin: pregabalin 150mg twice daily for 4 weeks
- Placebo First 4 Weeks: placebo and pregabalin given using a cross-over design
  pregabalin: pregabalin 150mg twice daily for 4 weeks
Period: Phase 1: Initial Intervention
Arm/Group | Pregabalin First 4 Weeks | Placebo First 4 Weeks
Started | 8 | 8
Completed | 0 | 0
Not Completed | 8 | 8
Not completed — Early study termination, poor enrollment | 8 | 8
Period: Phase 2: Cross Over
Arm/Group | Pregabalin First 4 Weeks | Placebo First 4 Weeks
Started | 0 | 0
Completed | 0 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No study analysis completed due to early termination due to poor enrollment
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin First 4 Weeks | Placebo First 4 Weeks | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.0 (8.9) | 36.3 (13.1) | 35.6 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 16
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Reduction in Average Pain Over the Last 7 Days of Each Arm Using an 11-point Scale (0-10)
Description: The primary objective of this protocol is to compare the reduction in pain using an 11-point scale (0-10) at four weeks of treatment. A responder will be defined as a subject noting a ≥50% reduction in pain using this scale.
  The NRS is an 11-point scale comprising a number from 0 through 10; 0 indicates "no pain", and 10 indicates the "worst imaginable pain".
  Outcomes measure not assessed due to early discontinuation because of poor recruitment. As such, the study was terminated prior to the designated follow up interval. Therefore, no outcomes data was collected.
Time Frame: 4 weeks
Population: Outcomes measure not assessed due to early discontinuation because of poor recruitment. As such, the study was terminated prior to the designated follow up interval. Therefore, no outcomes data was collected.
Arm/Group | Pregabalin/Placebo | Placebo/Pregabalin
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Effect on Anxiety and Depression in Women With Vulvodynia Based on the Kessler Psychological Distress Scale (K10)
Description: Subjects will complete the Kessler Psychological Distress Scale (K10). It is a measure of psychological distress. Scores will range from 10 to 50, with the higher the score, the higher the mental distress
  Data not measured due to early discontinuation of the study prior to the designated follow up time frame.
Time Frame: 4 weeks
Population: Data not measured due to early discontinuation of the study prior to the designated follow up time frame.
Arm/Group | Pregabalin First 4 Weeks | Placebo First 4 Weeks
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Description: Data not collected. Long term follow up not available for adverse events as study was discontinued early.
Arm/Group | Pregabalin/Placebo | Placebo/Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/8 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No